CLINICAL TRIAL: NCT03246737
Title: Premom: Pregnancy Remote Monitoring
Acronym: Premom
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Wilfried Gyselaers, prof. dr., Hasselt University
Other Study IDs: 14/078U
Record Dates: First submitted 2017-02-27; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Pregnancies, Cardiovascular Complications
MeSH Terms: conditions — Pregnancy Complications, Cardiovascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pregnant women
  Interventions: Other: monitoring

INTERVENTIONS:
Other: monitoring

SUMMARY:
Multiple cardiovascular adaptations happen during pregnancy. When gestational hypertensive disorders (GHD) occurs, these adaptations are abnormal. Approximately 5 - 8 % of all pregnant women develop GHD.

GHD is an pregnancy complication which is characterized by an elevated blood pressure (≥ 140/90 mm Hg) and sometimes the appearance of proteinuria (≥3 g/ 24 hours) after twenty weeks of pregnancy. When this remains uncured, GHD can have severe complications for both mother and child. For this reason, a close follow-up of women with a high risk for developing this condition is recommended. This to detect and threat GHD early.

Patients can be included when they are at least 10 weeks pregnant. Every pregnant women receives two devices to control daily here parameters in her home environment: a blood pressure monitor and an activity tracker. The women will be asked to perform two blood pressure measurements a day and to wear the activity tracker day and night. This data will be send by Bluetooth and Wi-Fi to the investigator in the hospital. Also will the women be asked to measure once a week her weight and send this to the hospital.

Name of the device Measurement Protocol Blood pressure monitor Blood pressure, heart rate Twice a day (morning and evening) Activity tracker Activity- and sleep pattern Day and night Weight scale (not remote) Weight Once a week (morning)

The investigator controls daily the incoming measurements and consults the responsible gyneacologist when events (= abnormal blood pressure or weight measurement) occurs. Depending on the decisions of the gyneacologist, following actions can be performed:

* Further observations
* Extra monitor
* Adjustments to the medication scheme
* Performing an 24 hours urine collection
* Admission to the prenatal observation ward When results are missing, the investigator contacts the women to ask of this measurement is due to personal or technical causes.

The purpose of this study part is to detect early signs of PE.

When patients gave birth, the data about the delivery (duration of labour, complications, mode of delivery, date of delivery, complications, parameters of the mother, specialties) and the neonate (gestational age, date and hour of birth, Apgar score, birth weight, length, complications and admission to the neonatal intensive care) will be collected. These data will be compared to the data of women who were admitted to the hospital for GHD, but who doesn't receive remote monitoring devices.

ELIGIBILITY:
Inclusion Criteria:

* > 10 weeks of gestation, in the possession of a Smartphone

Exclusion Criteria:

* congenital malformations of the fetus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
prenatal follow-up | up to 9 months (delivery)
  total number of prenatal appointments, monitors, echo's, prenatal hospitalizations, hospitalizations until delivery

SECONDARY OUTCOMES:
maternal hemodynamic outcomes | Day of delivery
  occurrence of essential hypertension/gestational hypertension/pre-eclampsie/help
birth weight | Day of delivery
  neonatal outcome
birth length | Day of delivery
  neonatal outcome
Apgar at 1' and 5' | Day of delivery
  neonatal outcome
admission to Neonatal Intensive Care | Day of delivery
  neonatal outcome

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Gyselaers, prof. dr., Principal Investigator — Hasselt University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lanssens D, Vandenberk T, Storms V, Thijs I, Grieten L, Bamelis L, Gyselaers W, Tang E, Luyten P. Changes in Intrapersonal Factors of Participants in the Pregnancy Remote Monitoring Study Who Are at Risk for Pregnancy-Induced Hypertension: Descriptive Quantitative Study. J Med Internet Res. 2023 Sep 6;25:e42686. doi: 10.2196/42686. PMID 37672324
- [Derived] Lanssens D, Vandenberk T, Lodewijckx J, Peeters T, Storms V, Thijs IM, Grieten L, Gyselaers W. Midwives', Obstetricians', and Recently Delivered Mothers' Perceptions of Remote Monitoring for Prenatal Care: Retrospective Survey. J Med Internet Res. 2019 Apr 15;21(4):e10887. doi: 10.2196/10887. PMID 30985286